CLINICAL TRIAL: NCT01505517
Title: Inspiratory Resistive Loading and Diaphragm Fatigue in Healthy Individuals and Individuals With Recurrent Low Back Pain
Brief Title: Inspiratory Resistive Loading and Diaphragm Fatigue
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Prof. dr. Simon Brumagne, KU Leuven
Other Study IDs: 2011_SBrumagne_DiaphFatigue; 1.5.104.03, G.0674.09 (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2012-07

CONDITIONS: Diaphragm Fatigue; Healthy; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- individuals with low back pain
- healthy controls

SUMMARY:
The aim of the study is to clarify whether specific loading of the inspiratory muscles induces contractile fatigue of the diaphragm muscle in healthy individuals and individuals with recurrent low back pain.

ELIGIBILITY:
Inclusion Criteria individuals with low back pain:

* Age: 18-35 years old
* At least 1 year of low back pain with/without referred pain in buttock/thigh
* At least 3 episodes of disabling low back pain
* At least a score of 20% on the Oswestry Disability Index
* Willingness to sign the informed consent

Inclusion Criteria healthy individuals:

* Age: 18-35 years old
* No history of low back pain
* A score of 0% on the Oswestry Disability Index
* Willingness to sign the informed consent

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson, multiple sclerosis, stroke, history of vestibular disorder, respiratory disease, pregnancy
* Radicular symptoms
* Not Dutch-speaking
* Strong opioids
* Neck pain
* Smoking history

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young flemish volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
transdiaphragmatic pressure | 18 months
  transdiaphragmatic pressure measurement in response to bilateral anterior magnetic phrenic nerve stimulation before and after an inspiratory resistive loading protocol

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, PhD, Principal Investigator — KU Leuven; Thierry Troosters, PhD, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

REFERENCES:
- [Background] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397
- [Background] Hermans G, Agten A, Testelmans D, Decramer M, Gayan-Ramirez G. Increased duration of mechanical ventilation is associated with decreased diaphragmatic force: a prospective observational study. Crit Care. 2010;14(4):R127. doi: 10.1186/cc9094. Epub 2010 Jul 1. PMID 20594319